CLINICAL TRIAL: NCT04083430
Title: Cytotoxicity of Yellow Fever Specific CD8 T Cells Following YF-17D Vaccination
Acronym: CYF-8
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YFV_001
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Cytotoxicity; Yellow Fever Vaccination Reaction
MeSH Terms: interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccine (Other): Yellow Fever Vaccine
  Interventions: Drug: Yellow Fever Vaccine

INTERVENTIONS:
Drug: Yellow Fever Vaccine — STAMARIL, powder and solvent for suspension for injection in pre-filled syringe.
  After reconstitution, 1 dose (0.5 ml) contains: Yellow fever virus1 17D-204 strain (live, attenuated) not less than 1000 IU.
  Powder and solvent for suspension for injection.
  Before reconstitution, the powder is homogeneous, beige to orange beige, and the solvent is a limpid solution.

SUMMARY:
Investigating cytotoxicity of yellow fever specific CD8 T cells following YF-17D vaccination and the following licensing of these epitope-specific CD8 T cells

DETAILED DESCRIPTION:
CD: cluster of differentiation YF: yellow fever

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years
* Informed consent given

Exclusion Criteria:

* Fever (orally >37,5 C) on day of vaccination
* Immunosuppressants
* Pregnant or breast feeding
* Severe immunodeficiency
* Known thymus dysfunction
* Allergy against egg
* Known haemophilia
* Previous severe reaction to vaccine
* Not willing to use anticonceptives 4 weeks after vaccination

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of cytotoxicity of the yellow fever specific (NS4B214LLWNGPMAV222) CD8 T cells 21(+/-3) days after vaccination with YF-17D | 21(+/-3) days
  Measured by flow cytometry
Incidence of cytotoxicity of the yellow fever specific (NS4B214LLWNGPMAV222) CD8 T cells 100 (+/- 40) days after vaccination with YF-17D | 100 (+/- 40) days
  Measured by flow cytometry

SECONDARY OUTCOMES:
% of patients with novel yellow fever vaccine epitopes according to HLA-type defining optimal timepoint for T cell licensing | 21(+/-3) days
  Measured by polymerase chain reaction
% of patients with novel yellow fever vaccine epitopes according to HLA-type defining optimal timepoint for T cell licensing | 100 (+/- 40) days
  Measured by polymerase chain reaction
Proportion of target cells killed ex vivo from in vivo generated YF-specific CD8+ T cells | 21(+/-3) days
  Measured by ex vivo killing assay
Proportion of target cells killed ex vivo from in vivo generated YF-specific CD8+ T cells | 100 (+/- 40) days
  Measured by ex vivo killing assay

CONTACTS AND LOCATIONS:
Overall Officials: Jesper D Gunst, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: We have developed an immunotherapy technology in which potent CTL responses are generated in vivo by vaccination and redirected to eliminate target cells using a bispecific Redirector of Vaccine-induced Effector Responses (RoVER) — https://pubmed.ncbi.nlm.nih.gov/37672868/